CLINICAL TRIAL: NCT07113405
Title: The Influence of Tea Extract on Maximal Voluntary Knee Contraction After 30 Minutes of Downhill Jogging: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Influence of Tea Extract on Maximal Voluntary Knee Contraction Following Downhill Jogging
Acronym: ITMVC-DJ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Fribourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2025-01302
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Muscle Recovery
Keywords: Protein; muscle recovery; Tea extract; EIMD
MeSH Terms: interventions — Proteins; Tea

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, placebo-controlled.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Protein and tea extract (Experimental): This group will receive a recovery drink containing protein and tea extract.
  Interventions: Dietary Supplement: Protein and tea extract
- Protein (Active Comparator): This group will receive a recovery drink containing protein without tea extract.
  Interventions: Dietary Supplement: Protein
- Placebo (Placebo Comparator): This group will receive a recovery drink containing a placebo product. The placebo product is a non-isoenergetic, non-protein, artificially flavoured liquid.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Protein and tea extract — Participants in this group will receive 4 times a recovery drink containing protein and tea extract.
  Arms: Protein and tea extract
Dietary Supplement: Protein — Participants of this group will receive ten times a recovery drink containing only protein without tea extract.
  Arms: Protein
Dietary Supplement: Placebo — Participants of this group will receive 10 times a placebo containing no protein nor tea extract.
  Arms: Placebo

SUMMARY:
In this research project, we want to investigate whether the combined intake of proteins and tea extract has an influence on muscle regeneration compared to the sole intake of proteins or a placebo product. In the study, you will be randomly assigned to one of 3 groups. Neither the research group nor you will know which group you are assigned to. The study lasts 5 days for you as a participant. During these 5 days you will have to attend a total of 5 appointments in our laboratory. The groups differ only in the intake of the regeneration product, otherwise all measurements and appointments are identical. You will jog downhill for 30 minutes on the first day in order to strain your muscles. In order to be able to draw conclusions about the regeneration of your muscles, we will carry out the following measurements on all 5 days: Blood sampling at the fingertip, ultrasound of the thigh muscle, pain tolerance of the thigh muscle, strength tests of the thigh muscle, muscle function of the thigh muscle and jumping performance.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged between 18-40 years
* Healthy subjects

Exclusion Criteria:

* Any type of food allergy (e.g. nuts)
* Health-related problems according to the "Physical Activity Readiness Questionnaire (PAR-Q)
* Current injury of the lower extremities
* Serious clinical back pain or current back injuries
* Orthopedic disorders
* Cardiovascular diseases
* Current Intake of blood-thinning medication
* Current Intake of anti-inflammatory medication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in maximum knee extension force immediately after training-induced muscle damage and 24, 48, 72, and 96 hours thereafter compared to baseline. | 5 days
  The maximal force is measured in Nm while the participant is seated on an isokinetic device.
Change in jump performance immediately after training-induced muscle damage and 24, 48, 72, and 96 hours thereafter compared to baseline. | 5 days
  The jump performance is measured in cm while the participant are performing counter movement jumps.
Change in perceived pain immediately after training-induced muscle damage and 24, 48, 72, and 96 hours thereafter compared to baseline. | 5 days
  Perceived pain is measured in Pa while the participant is seated on the isokinetic device. The measurement point is on vastus medialis muscle.
Change in muscle thickness immediately after training-induced muscle damage and 24, 48, 72, and 96 hours thereafter compared to baseline. | 5 days
  Muscle thickness is measured with b-mode ultrasound in mm while the participant is sitting on the isokinetic device. The measurement point is on the vastus medialis muscle.
Change in creatine kinase levels immediately after exercise-induced muscle damage and 24, 48, 72, and 96 hours thereafter compared to baseline. | 5 days
  Creatine kinase is measured in U/L and determined using a capillary finger blood sample of 0.25 ml.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Fribourg, Fribourg, Canton of Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No
It is planned that only our research group will analyze and publish the data. Therefore, the data will not be passed on to other researchers.

REFERENCES:
- [Result] Volpe-Fix AR, de Franca E, Silvestre JC, Thomatieli-Santos RV. The Use of Some Polyphenols in the Modulation of Muscle Damage and Inflammation Induced by Physical Exercise: A Review. Foods. 2023 Feb 21;12(5):916. doi: 10.3390/foods12050916. PMID 36900433
- [Result] Isaacs AW, Macaluso F, Smith C, Myburgh KH. C-Reactive Protein Is Elevated Only in High Creatine Kinase Responders to Muscle Damaging Exercise. Front Physiol. 2019 Feb 11;10:86. doi: 10.3389/fphys.2019.00086. eCollection 2019. PMID 30804809
- [Result] Hug F, Avrillon S, Del Vecchio A, Casolo A, Ibanez J, Nuccio S, Rossato J, Holobar A, Farina D. Analysis of motor unit spike trains estimated from high-density surface electromyography is highly reliable across operators. J Electromyogr Kinesiol. 2021 Jun;58:102548. doi: 10.1016/j.jelekin.2021.102548. Epub 2021 Mar 30. PMID 33838590
- [Result] Fischer AA. Pressure algometry over normal muscles. Standard values, validity and reproducibility of pressure threshold. Pain. 1987 Jul;30(1):115-126. doi: 10.1016/0304-3959(87)90089-3. PMID 3614975
- [Result] Del Vecchio A, Casolo A, Negro F, Scorcelletti M, Bazzucchi I, Enoka R, Felici F, Farina D. The increase in muscle force after 4 weeks of strength training is mediated by adaptations in motor unit recruitment and rate coding. J Physiol. 2019 Apr;597(7):1873-1887. doi: 10.1113/JP277250. Epub 2019 Feb 6. PMID 30727028
- [Result] Coratella G, Varesco G, Rozand V, Cuinet B, Sansoni V, Lombardi G, Vernillo G, Mourot L. Downhill running increases markers of muscle damage and impairs the maximal voluntary force production as well as the late phase of the rate of voluntary force development. Eur J Appl Physiol. 2024 Jun;124(6):1875-1883. doi: 10.1007/s00421-023-05412-z. Epub 2024 Jan 10. PMID 38195943
- [Result] Botter A, Vieira TM, Loram ID, Merletti R, Hodson-Tole EF. A novel system of electrodes transparent to ultrasound for simultaneous detection of myoelectric activity and B-mode ultrasound images of skeletal muscles. J Appl Physiol (1985). 2013 Oct 15;115(8):1203-14. doi: 10.1152/japplphysiol.00090.2013. Epub 2013 Aug 1. PMID 23908313